CLINICAL TRIAL: NCT06203262
Title: A Pre-Market, First-In-Human, Pilot, Interventional, Clinical Investigation to Evaluate Safety and Feasibility of the FieldForce™ Ablation System in Symptomatic Patients With Ventricular Arrhythmia
Brief Title: Ventricular Catheter Ablation Study (VCAS)
Acronym: VCAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Field Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FM-PFA-VT-2023
Record Dates: First submitted 2023-12-30; First posted 2024-01-12 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Ventricular Tachyarrhythmia; Ventricular Arrythmia; PVC - Premature Ventricular Complex; PVC - Premature Ventricular Contraction; Ventricular Tachycardia
Keywords: ventricular tachycardia; VT; premature ventricular contractions; PVC; electroporation; pulse field ablation; PFA
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Premature Complexes | interventions — Irreversible Electroporation Therapy

STUDY DESIGN:
Intervention Model Description: Prospective single arm safety and feasibility study. There are two populations that will be enrolled and analyzed separately: patients being treated for ventricular tachycardia (VCAS-I) and patients with frequent premature ventricular contractions (VCAS-II). The intervention in both cases is similar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Ventricular Tachycardia (VCAS-I) (Experimental): Patients with ventricular tachycardia meeting class II-a/b indications in European guideline for catheter ablation, with a clinical VT event detected by an implanted ICD
  Interventions: Device: FieldForce™ Ablation System Ventricular Tachycardia
- Premature Ventricular Contractions (VCAS-II) (Experimental): For VCAS-II group, patients with symptomatic frequent unifocal premature ventricular complexes (PVCs) meeting class II-a/b indications based on European guidelines for catheter ablation. For VCAS-II, documentation of frequent PVCs by 24 hours Holter with >15% PVC burden for asymptomatic patients and >5% PVC burden for symptomatic patients within the last 60 days.
  Interventions: Device: FieldForce™ Ablation System Premature Ventricular Contractions

INTERVENTIONS:
Device: FieldForce™ Ablation System Ventricular Tachycardia — Catheter ablation is a minimally invasive procedure. The physician advances multiple catheters into the heart that are used to diagnose and localize abnormal cardiac tissue involved in the initiation and maintenance of ventricular tachycardia and/or PVCs. Once the abnormal tissue is identified a specialized catheter is advanced to the target and energy is applied to destroy the abnormal tissue. The intervention will be identical to the conventional procedure except that an investigational ablation catheter will be used to deliver energy.
  Other Names: Pulse Field Ablation
  Arms: Ventricular Tachycardia (VCAS-I)
Device: FieldForce™ Ablation System Premature Ventricular Contractions — Catheter ablation is a minimally invasive procedure. The physician advances multiple catheters into the heart that are used to diagnose and localize abnormal cardiac tissue involved in the initiation and maintenance of ventricular tachycardia and/or PVCs. Once the abnormal tissue is identified a specialized catheter is advanced to the target and energy is applied to destroy the abnormal tissue. The intervention will be identical to the conventional procedure except that an investigational ablation catheter will be used to deliver energy.
  Other Names: Pulse Field Ablation
  Arms: Premature Ventricular Contractions (VCAS-II)

SUMMARY:
This is a prospective safety and feasibility study to evaluate the safety of the FieldForce™ Ablation system in patients with ventricular arrhythmia divided into two groups: VT (VCAS-I) and frequent premature ventricular complex (VCAS-II).

DETAILED DESCRIPTION:
Summary:

Ventricular arrythmias are common but often undertreated. The most effective pharmacologic management and implantable devices are used to treat deadly arrythmias like ventricular tachycardia (VT) and ventricular fibrillation (VF). However, the efficacy of antiarrhythmic drugs (AADs) has been proven to be low, and implantable cardioverter defibrillators (ICDs) treat VT but do not prevent it. Prospective trials demonstrate that VT ablation is by far the most effective therapy for ventricular tachycardia and in some cases it is curative. Despite overwhelming evidence that catheter ablation is superior, there are many technical barriers that prevent widespread application of this therapy. Furthermore, non-fatal ventricular arrythmias such as premature ventricular contractions (PVCs) are treatable by catheter ablation. The technical challenges facing VT and PVC ablations are similar as current technologies are optimized to treat atrial arrythmias often at the expense of performance in the ventricle.

Pulsed field ablation (PFA) is a new ablation method for the therapy of arrhythmias. PFA is considered as a non-thermal and low-energy method of ablation. This technique is characterized by pulse trains of short-duration and high-voltage electrical impulses that result in electric field-mediated tissue injury. The very strong electric fields put strain on cellular compartmentalization. These changes can be reversible, and cells can recover with no consequences; however, if compartmentalization is disrupted for an extended period of time, it results in metabolic injury and cell death. This mechanism is also known as electroporation. Different cell types are sensitive to these types of insults leading to tissue selectivity in the heart. Clinical studies have already demonstrated the feasibility and safety of PFA for the treatment of atrial fibrillation. However, there is less data on the application of PFA for VT.

Therefore, this Pre-Market, First-In-Human, Pilot, Interventional, Clinical Investigation aims to evaluate Safety and Feasibility of the FieldForce™ Ablation system in patients with ventricular tachycardia divided into two groups: ventricular tachycardia (VCAS-I) and unifocal premature ventricular complex (VCAS-II).

ELIGIBILITY:
INCLUSION:

1. Signed patient informed consent form (ICF).
2. Female and male participants between 18 and 80 years.
3. For VCAS-I group, patients with VT meeting class II-a/b indications in European guideline for catheter ablation, with a clinical VT event detected by an implanted ICD
4. For VCAS-II group, patients with frequent premature ventricular complexes (PVCs) meeting class II-a/b indications based on European guidelines for catheter ablation.
5. For VCAS-II, documentation of frequent PVCs by 24 hours Holter with >15% PVC burden for asymptomatic patients and >5% PVC burden for symptomatic patients within the last 60 days.

EXCLUSION:

1. Body Mass Index > 40.
2. Pacemaker dependence.
3. Ineligible for ablation according to Physician judgement (including but not limited to known to have protruding left ventricular thrombus or have implanted mechanical aortic and mitral valves).
4. Recent MI (less than 90 days) or another reversible cause of VT (e.g., electrolyte abnormalities, drug-induced arrhythmia).
5. The presence of inferior vena cava embolic protection filter devices.
6. Recent cardiac surgery (less than 2 months)
7. NYHA Class IV.
8. Hemodynamically severe valvular disease that precludes ablation. Severity will be evaluated by using echocardiography, according to AHA and European guidelines.
9. Uncontrolled abnormal bleeding and/or clotting disorder.
10. Contraindication to systemic or oral anticoagulation.
11. Serious or untreated medical conditions that would prevent participation in the study, interfere with assessment or therapy, or confound data or its interpretation, including but not limited to solid organ or hematologic transplant, or currently being evaluated for an organ transplant.
12. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or significant dyspnea.
13. Chronic renal insufficiency of eGFR< 30 mL/min/1.73 m2.
14. Active malignancy
15. Untreated clinically significant infection.
16. Life expectancy is less than one year.
17. Clinically significant psychological condition that in the investigator's opinion would prohibit the subject's ability to meet the study requirements.
18. Prohibitively distorted cardiac anatomy due to congenital heart disease.
19. Had a recent percutaneous coronary intervention (<1 month).
20. Participation in another investigational study or treatment with any investigational drug within the previous 30 days that would interfere with this study.
21. Patient is not able to understand the nature of this study or is unwilling or unable to attend the study procedures.
22. Pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-04-12 (Estimated); Study Completion 2025-04-12 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint Acute | < 30 days
  device-related or procedure-related Serious Adverse Events

SECONDARY OUTCOMES:
Reduction in clinical arrhythmia burden (VCAS-I) | baseline, 90 days & 180 days
  Compare the baseline arrhythmia logs recorded on the ICD to post procedure arrhythmia logs
Reduction in clinical arrhythmia burden (VCAS-II) | baseline, after 90 days and no longer than 120 days
  Compare the baseline 24-hour Holter PVC burden after ablation
Procedure duration (average minutes of procedure time) | 1 day
  Time points in the procedure will be recorded and stratified by group
Evaluate VT inducibility (VCAS-I) pre and post ablation | index procedure
  VT inducibility using programed stimulation using two drive cycle lengths and triple extra stimuli will be performed.
Detect Ischemic scar homogenization (VCAS-I) | baseline and 90 days
  Ischemic scar homogenization using cardiac magnetic resonance (CMR) will be performed before ablation at baseline and 90 days.

OTHER OUTCOMES:
Device Deficiencies | 180 days
  Device deficiencies/incidents before, during and after the use of the device.
Adverse Events and Serious Adverse Events | 180 days
  Adverse events and serious adverse events unrelated to study device or procedure over the duration of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Na Homolce Hospital, Prague
  - IKEM, Prague

REFERENCES:
- [Derived] Reddy VY, Koruth JS, Peichl P, Petru J, Funasako M, Skoda J, Watanabe K, Nies M, Kautzner J, Neuzil P. High-Voltage Focal Pulsed Field Ablation to Treat Scar-Related Ventricular Tachycardia: The First-in-Human VCAS Trial. Circulation. 2025 Dec 16;152(24):1691-1704. doi: 10.1161/CIRCULATIONAHA.125.077025. Epub 2025 Oct 10. PMID 41071961